CLINICAL TRIAL: NCT03319381
Title: Implementation of New Standard Operating Procedures for Geriatric Trauma Patients With Multiple Injuries
Brief Title: Geriatric Polytrauma SOP
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: USZ-TRA-SPRKA001
Record Dates: First submitted 2017-10-17; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Geriatrics
Keywords: Algorithm; In-hospital mortality; Multiple trauma; Standard of care
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- w/o SOP: Time period 1: 2000-2006, without new SOPs
  Interventions: Behavioral: Following new SOPs
- SOP: Time period 2: 2010-2012, after implementation of the new SOPs
  Interventions: Behavioral: Following new SOPs

INTERVENTIONS:
Behavioral: Following new SOPs — The new SOPs comprised early whole-body CT, damage control surgery, and the use of goal-directed coagulation management and are based on the ATLS® concept, which was the strictly followed protocol before implementation of the new SOPs

SUMMARY:
This study investigated whether there were improvements in the in-hospital mortality, infection rate, and rate of palliative care among geriatric trauma patients after the implementation of new standard operating procedures (SOPs) for the resuscitation room. These new SOPs, comprising early whole-body computed tomography (CT), damage control surgery, and the use of goal-directed coagulation management, were designed for severely injured adult trauma patients

DETAILED DESCRIPTION:
This study involved the analysis of a prospective single-centre database. Patients admitted via the resuscitation room with need for intensive care treatment after the resuscitation room phase were included and compared before the implementation of the new SOPs (between 1 January, 2000 and 31 December, 2006) and after their implementation in 2009 (between 1 January, 2010 and 31 December, 2012) of our level-I trauma centre.

ELIGIBILITY:
Inclusion Criteria:

Inclusion in internal trauma database

Exclusion Criteria:

Comprised age < 65 years, ISS < 9, and transfers from other hospitals.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Trauma patients admitted via the resuscitation room with need for intensive care treatment after the resuscitation room phase were included in the internal trauma database
Sampling Method: Non-Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | 30 days
  In-hospital mortality

SECONDARY OUTCOMES:
Infections | 30 days
  Infections
Rate of palliative care | 30 days
  Rate of palliative care

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peterer L, Ossendorf C, Jensen KO, Osterhoff G, Mica L, Seifert B, Werner CML, Simmen HP, Pape HC, Sprengel K. Implementation of new standard operating procedures for geriatric trauma patients with multiple injuries: a single level I trauma centre study. BMC Geriatr. 2019 Dec 19;19(1):359. doi: 10.1186/s12877-019-1380-z. PMID 31856739